CLINICAL TRIAL: NCT03587207
Title: Immunogenicity and Safety of Meningococcal MenABCWY Vaccine, and of rMenB+OMV NZ and MenACWY Administered Concomitantly in the Same Arm or in 2 Different Arms, or Alone
Brief Title: Study to Assess Potential Immune Interference When GlaxoSmithKline (GSK) Biologicals' MenABCWY Vaccine is Administered to Healthy Subjects Aged 10-25 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 208205; 2017-005128-12 (EudraCT Number)
Record Dates: First submitted 2018-06-29; First posted 2018-07-16 (Actual); Results first posted 2020-01-02 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-01

CONDITIONS: Meningitis, Meningococcal
Keywords: Meningitis; Concomitantly; Adolescent; Neisseria meningitidis; Healthy subjects; Adult
MeSH Terms: conditions — Meningitis, Meningococcal; Meningitis | interventions — 4CMenB vaccine; Vaccines; MenACWY; Meningococcal Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- MenABCWY Group (Experimental): Healthy subjects between, and including, 10 to 25 years of age at the time of the first vaccination (equally distributed across the 2 age strata of 10 to 17 years and 18 to 25 years) received one dose of MenABCWY twice, 2 months apart (Day 1 and Day 61).
  Interventions: Biological: MenABCWY vaccine
- rMenBOMV+ACWY_S Group (Active Comparator): Healthy subjects between, and including, 10 to 25 years of age at the time of the first vaccination (equally distributed across the 2 age strata of 10 to 17 years and 18 to 25 years) concomitantly received one dose of rMenB+OMV NZ (Bexsero) and one dose of MenACWY (Menveo) in the same arm twice, 2 months apart (Day 1 and Day 61).
  Interventions: Biological: rMenB+OMV NZ (Bexsero) vaccine; Biological: MenACWY (Menveo) vaccine
- rMenBOMV+ACWY_D Group (Active Comparator): Healthy subjects between, and including, 10 to 25 years of age at the time of the first vaccination (equally distributed across the 2 age strata of 10 to 17 years and 18 to 25 years) concomitantly received one dose of rMenB+OMV NZ (Bexsero) and one dose of MenACWY (Menveo) in 2 different arms twice, 2 months apart (Day 1 and Day 61).
  Interventions: Biological: rMenB+OMV NZ (Bexsero) vaccine; Biological: MenACWY (Menveo) vaccine
- rMenBOMV Group (Active Comparator): Healthy subjects between, and including, 10 to 25 years of age at the time of the first vaccination (equally distributed across the 2 age strata of 10 to 17 years and 18 to 25 years) received one dose of rMenB+OMV NZ (Bexsero) twice, 2 months apart (Day 1 and Day 61).
  Interventions: Biological: rMenB+OMV NZ (Bexsero) vaccine
- MenACWY Group (Active Comparator): Healthy subjects between, and including, 10 to 25 years of age at the time of the first vaccination (equally distributed across the 2 age strata of 10 to 17 years and 18 to 25 years) received one dose of MenACWY (Menveo) once at Day 1, which was the first and last vaccination for MenACWY group.
  Interventions: Biological: MenACWY (Menveo) vaccine

INTERVENTIONS:
Biological: MenABCWY vaccine — Two doses administered intramuscularly in the deltoid region of the non-dominant arm.
  Arms: MenABCWY Group
Biological: rMenB+OMV NZ (Bexsero) vaccine — Two doses administered 2 months apart intramuscularly in the deltoid region of the non-dominant arm to subjects randomised to the rMenBOMV+ACWY_S Group, rMenBOMV+ACWY_D Group and rMenBOMV Group
  Arms: rMenBOMV Group; rMenBOMV+ACWY_D Group; rMenBOMV+ACWY_S Group
Biological: MenACWY (Menveo) vaccine — Two doses administered intramuscularly in the deltoid region of the dominant/non-dominant arm to subjects randomised to the rMenBOMV+ACWY_S Group and rMenBOMV+ACWY_D Group and one dose administered intramuscularly in the deltoid region of the dominant/non-dominant arm to subjects randomised to the MenACWY Group
  Arms: MenACWY Group; rMenBOMV+ACWY_D Group; rMenBOMV+ACWY_S Group

SUMMARY:
The purpose of the current study is to evaluate whether there is immune interference when MenABCWY [consisting of MenACWY lyophilized component and rMenB+OMV NZ (Bexsero) liquid component] is administered to healthy adolescents and adults following a 2-dose vaccination schedule with MenABCWY administered 2 months apart.

ELIGIBILITY:
Inclusion Criteria:

* Subjects and/or subjects' parent(s)/Legally Acceptable Representative(s) (LARs) who, in the opinion of the investigator, can and will comply, with the requirements of the protocol (e.g. completion of the paper diary (pDiary), return for follow-up visits, availability for all visits scheduled in the study).
* Written informed consent obtained from the subject and/or from the parent(s)/LAR(s) of the subject prior to performing any study specific procedure.
* Written informed assent obtained from subjects below the legal age of consent prior to performing any study specific procedure.
* A male or female between, and including, 10 to 25 years of age at the time of the first vaccination.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre menarche, current bilateral tubal ligation or occlusion, hysterectomy, or bilateral ovariectomy.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced highly effective contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue highly effective contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Female planning to become pregnant or planning to discontinue contraceptive precautions
* Pregnant or lactating female
* Child in care
* Current or previous, confirmed or suspected disease caused by N. meningitidis.
* Known contact to an individual with any laboratory confirmed N. meningitidis infection within 60 days prior to enrolment.
* Previous vaccination against N. meningitidis at any time prior to informed consent.
* Progressive, unstable or uncontrolled clinical conditions.
* Hypersensitivity, including allergy, to any component of vaccines, medicinal products or medical equipment whose use is foreseen in this study.
* Clinical conditions representing a contraindication to IM vaccination and blood draws.
* Abnormal function of the immune system resulting from:

  * Clinical conditions.
  * Systemic administration of corticosteroids (oral/intravenous/IM) for more than 14 consecutive days within 90 days prior to informed consent.
  * Administration of antineoplastic and immune modulating agents or radiotherapy within 90 days prior to informed consent.
* Received immunoglobulins or any blood products within 180 days prior to informed consent.
* Received an investigational or non registered medicinal product within 30 days prior to informed consent.
* Any other clinical condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subject due to participation in the study.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non investigational vaccine/product.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by physical examination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Are obese at screening.
* Family history of congenital or hereditary immunodeficiency.
* History of neuroinflammatory or autoimmune condition.
* History of significant neurological disorder or seizure.
* Serious chronic illness.
* History of chronic alcohol consumption and/or drug abuse.
* Any study personnel as an immediate family or household member.
* Administration of a vaccine not foreseen by the study protocol in the period starting 14 days (for inactivated vaccines), 28 days (for live vaccines), or 7 days (for influenza vaccines) before each dose and ending 14 days (for inactivated vaccines), 28 days (for live vaccines), or 7 days (for influenza vaccines) after each dose of study vaccine(s) administration.
* Thrombocytopenia, bleeding disorders, or be receiving anticoagulant therapy.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 520 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Beran J, Drazan D, Enweonye I, Bhusal C, Toneatto D. Immunogenicity and Safety of Investigational MenABCWY Vaccine and of 4CMenB and MenACWY Vaccines Administered Concomitantly or Alone: a Phase 2 Randomized Study of Adolescents and Young Adults. mSphere. 2021 Dec 22;6(6):e0055321. doi: 10.1128/mSphere.00553-21. Epub 2021 Nov 17. PMID 34787449

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 1 center at Czechia.
Pre-assignment Details: Out of the total 520 subjects enrolled in this study, 500 subjects received the vaccination. Among the 20 subjects that were not vaccinated, 15 did not fuflill eligibility criteria and 5 were excluded due to other reasons.
Period: Overall Study
Arm/Group | MenABCWY Group | rMenBOMV+ACWY_S Group | rMenBOMV+ACWY_D Group | rMenBOMV Group | MenACWY Group
Started | 100 | 104 | 100 | 94 | 102
Completed | 100 | 104 | 100 | 94 | 102
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MenABCWY Group | rMenBOMV+ACWY_S Group | rMenBOMV+ACWY_D Group | rMenBOMV Group | MenACWY Group | Total
Number analyzed (Participants) | 100 | 104 | 100 | 94 | 102 | 500
Age, Continuous [Mean (Standard Deviation); unit: Years] | 17.1 (4.34) | 16.9 (4.28) | 17.1 (4.49) | 17.4 (4.64) | 17.1 (4.57) | 17.1 (4.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 48 | 49 | 53 | 49 | 246
  Male | 53 | 56 | 51 | 41 | 53 | 254
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: WHITE | 100 | 104 | 100 | 94 | 102 | 500

OUTCOME MEASURES:

1. Primary Outcome: Human Serum Bactericidal Activity (hSBA) Adjusted Geometric Mean Titers (GMTs) Against All of N. Meningitidis Serogroup B Test Strains (Pooled), One Month After Last Vaccination.
Description: hSBA titers against all of N. meningitidis serogroup B test strains were calculated in terms of GMTs. Serogroup B strains tested were M14459 (factor H binding protein; fHbp), 96217 (Neisserial adhesin A; NadA), NZ98/254 (PorA), and M070241084 (Neisseria heparin binding antigen; NHBA). The serogroup B strains were grouped together to perform a pooled analysis. Adjusted means were obtained from ANCOVA model fitted to all of the Serogroup B test strains, study group, test strain and center as fixed effects; zero-centered pre-vaccination log-transformed titer was included as a continuous covariate.
Time Frame: 1 month after last vaccination i.e.: at Day 91 for all groups except for the MenACWY Group
Population: Analysis performed on Per Protocol Set(PPS) for immunogenicity that included subjects without major protocol violations & whose assay results were available for atleast 1 serogroup/B strain at Day 91 for all study groups except MenACWY group that was not considered for this analysis as only serogroup B strains were assessed in this outcome measure
Measure: Geometric Mean (80% Confidence Interval); unit: titers
Arm/Group | MenABCWY Group | rMenBOMV+ACWY_S Group | rMenBOMV+ACWY_D Group | rMenBOMV Group
Number analyzed (Participants) | 98 | 100 | 97 | 90
titers | 31.84 [28.18 to 35.98] | 38.48 [34.23 to 43.26] | 40.08 [35.44 to 45.33] | 42.38 [37.31 to 48.13]
Statistical Analysis 1: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV+ACWY_D Group; Immune interference due to stress to lymph nodes (lymph-node effect) in rMenBOMV+ACWY_S versus rMenBOMV+ACWY_D study groups, on the pooled B strains, one month after last vaccination; Test type: Other — rMenBOMV+ACWY_S is to be declared statistically inferior if the 2-sided 80% CIs of the between group ratio of the GMT with rMenBOMV+ACWY_D as control is lower than 1 at 1 month after last vaccination. The following ANCOVA model is used: fixed-effect model including age strata, study group, strain and center as fixed effects. The pre vaccination (Baseline) log-transformed titer with centering at zero is included as a continuous covariate; ANCOVA; An interaction between strain and pre-vaccination log transformed titer is included in the model to fit to the serogroup B test strain data only; Geometric mean ratio = 0.96, 80% CI 2-sided [0.83 to 1.10]

2. Primary Outcome: hSBA Adjusted GMTs Against Each of the N. Meningitidis Serogroup B Test Strains and N. Meningitidis Serogroups A, C, W-135, and Y, One Month After Last Vaccination.
Description: hSBA titers against each of the N. meningitidis serogroup B test strains and N. meningitidis serogroups A, C, W-135, and Y were calculated in terms of GMTs. Serogroup B strains tested were M14459 (factor H binding protein; fHbp), 96217 (Neisserial adhesin A; NadA), NZ98/254 (PorA), and M070241084 (Neisseria heparin binding antigen; NHBA). Adjusted means were obtained from ANCOVA model fitted to each Serogroup (Strain) individually, study group and center as fixed effects and zero-centered pre-vaccination log-transformed titer as a continuous covariate.
Time Frame: 1 month after last vaccination i.e.: at Day 91 for all groups except the MenACWY Group, and at Day 31 for the MenACWY Group.
Population: Analysis was performed on PPS for immunogenicity that included subjects who had no major protocol violations and whose assay results were available for at least 1 serogroup or B strain at Day 91 for all study groups except MenACWY Group or at Day 31 for the MenACWY Group.
Measure: Geometric Mean (80% Confidence Interval); unit: titers
Arm/Group | MenABCWY Group | rMenBOMV+ACWY_S Group | rMenBOMV+ACWY_D Group | rMenBOMV Group | MenACWY Group
Number analyzed (Participants) | 98 | 101 | 97 | 90 | 97
titers
  Meningitis B M14459 (fHbp): number analyzed (Participants) | 97 | 100 | 96 | 90 | 97
  Meningitis B M14459 (fHbp) | 23.91 [20.52 to 27.86] | 23.34 [20.16 to 27.01] | 23.23 [19.91 to 27.10] | 22.87 [19.52 to 26.80] | 2.48 [2.13 to 2.89]
  Meningitis B 96217(NadA): number analyzed (Participants) | 98 | 100 | 97 | 90 | 96
  Meningitis B 96217(NadA) | 81.09 [69.24 to 94.97] | 102.68 [88.24 to 119.50] | 97.54 [83.18 to 114.39] | 113.54 [96.25 to 133.93] | 4.15 [3.54 to 4.86]
  Meningitis B NZ98/254(PorA): number analyzed (Participants) | 98 | 100 | 97 | 89 | 97
  Meningitis B NZ98/254(PorA) | 12.97 [10.89 to 15.45] | 16.39 [13.86 to 19.39] | 21.12 [17.71 to 25.18] | 20.97 [17.47 to 25.16] | 2.15 [1.81 to 2.57]
  Meningitis B M07-0241084(NHBA): number analyzed (Participants) | 98 | 100 | 96 | 89 | 95
  Meningitis B M07-0241084(NHBA) | 13.08 [11.09 to 15.43] | 18.00 [15.35 to 21.11] | 22.59 [19.12 to 26.69] | 25.34 [21.30 to 30.13] | 4.08 [3.45 to 4.82]
  Meningitis A: number analyzed (Participants) | 97 | 101 | 97 | 90 | 93
  Meningitis A | 104.90 [87.02 to 126.47] | 187.52 [156.94 to 224.05] | 204.01 [169.06 to 246.18] | 94.91 [78.26 to 115.12] | 52.03 [43.01 to 62.95]
  Meningitis C: number analyzed (Participants) | 98 | 100 | 97 | 90 | 97
  Meningitis C | 172.99 [140.43 to 213.09] | 144.80 [118.48 to 176.97] | 145.42 [117.91 to 179.34] | 32.01 [25.75 to 39.79] | 34.66 [28.09 to 42.78]
  Meningitis W: number analyzed (Participants) | 98 | 100 | 96 | 90 | 97
  Meningitis W | 260.11 [219.31 to 308.51] | 245.63 [208.40 to 289.52] | 254.20 [213.76 to 302.30] | 193.58 [161.68 to 231.76] | 80.11 [67.42 to 95.19]
  Meningitis Y: number analyzed (Participants) | 97 | 100 | 97 | 89 | 96
  Meningitis Y | 219.52 [173.10 to 278.39] | 186.08 [148.25 to 233.55] | 204.92 [161.40 to 260.16] | 3.66 [2.86 to 4.69] | 92.41 [72.75 to 117.37]
Statistical Analysis 1: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV+ACWY_D Group; Immune interference due to stress to lymph nodes (lymph-node effect) in rMenBOMV+ACWY_S versus rMenBOMV+ACWY_D study groups, on the Meningitis B M14459 (fHbp) strain, one month after last vaccination; Test type: Other — M14459 strain-Between group ratios for comparison of rMenBOMV+ACWY_S and rMenBOMV+ACWY_D groups; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 1.00, 80% CI 2-sided [0.84 to 1.20]
Statistical Analysis 2: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV+ACWY_D Group; Immune interference due to stress to lymph nodes (lymph-node effect) in rMenBOMV+ACWY_S versus rMenBOMV+ACWY_D study groups, on the Meningitis B 96217 (NadA) strain, one month after last vaccination; Test type: Other — 96217 strain-Between group ratios for comparison of rMenBOMV+ACWY_S and rMenBOMV+ACWY_D groups; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 1.05, 80% CI [0.88 to 1.26]
Statistical Analysis 3: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV+ACWY_D Group; Immune interference due to stress to lymph nodes (lymph-node effect) in rMenBOMV+ACWY_S versus rMenBOMV+ACWY_D study groups, on the Meningitis B NZ98/254 (PorA) strain, one month after last vaccination; Test type: Other — NZ98/254 strain-Between group ratios for comparison of rMenBOMV+ACWY_S and rMenBOMV+ACWY_D groups; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.78, 80% CI 2-sided [0.64 to 0.95]
Statistical Analysis 4: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV+ACWY_D Group; Immune interference due to stress to lymph nodes (lymph-node effect) in rMenBOMV+ACWY_S versus rMenBOMV+ACWY_D study groups, on the Meningitis B M07-0241084 (NHBA) strain, one month after last vaccination; Test type: Other — M07-0241084 strain- Between group ratios for comparison of rMenBOMV_ACWY_S group and rMenBOMV+ACWY_D group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.80, 80% CI 2-sided [0.66 to 0.96]
Statistical Analysis 5: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV+ACWY_D Group; Immune interference due to stress to lymph nodes (lymph-node effect) in rMenBOMV+ACWY_S versus rMenBOMV+ACWY_D study groups, on the Meningitis serogroup A, one month after last vaccination; Test type: Other — Serogroup A- Between group ratio for comparison of rMenBOMV+ACWY_S group and rMenBOMV+ACWY_D group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.92, 80% CI 2-sided [0.74 to 1.14]
Statistical Analysis 6: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV+ACWY_D Group; Immune interference due to stress to lymph nodes (lymph-node effect) in rMenBOMV+ACWY_S versus rMenBOMV+ACWY_D study groups, on the Meningitis serogroup C, one month after last vaccination; Test type: Other — Serogroup C- Between group ratio for comparison of rMenBOMV+ACWY_S group and rMenBOMV+ACWY_D group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 1.00, 80% CI 2-sided [0.78 to 1.27]
Statistical Analysis 7: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV+ACWY_D Group; Immune interference due to stress to lymph nodes (lymph-node effect) in rMenBOMV+ACWY_S versus rMenBOMV+ACWY_D study groups, on the Meningitis serogroup W, one month after last vaccination; Test type: Other — Serogroup W- Between group ratios for comparison of rMenBOMV+ACWY_S group and rMenBOMV+ACWY_D group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.97, 80% CI 2-sided [0.79 to 1.18]
Statistical Analysis 8: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV+ACWY_D Group; Immune interference due to stress to lymph nodes (lymph-node effect) in rMenBOMV+ACWY_S versus rMenBOMV+ACWY_D study groups, on the Meningitis serogroup Y, one month after last vaccination; Test type: Other — Serogroup Y- Between group ratio for comparison of rMenBOMV+ACWY_S group and rMenBOMV+ACWY_D group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.91, 80% CI 2-sided [0.69 to 1.19]
Statistical Analysis 9: Comparison: MenABCWY Group vs rMenBOMV+ACWY_S Group; Other unknown interference in MenABCWY versus rMenBOMV+ACWY_S study groups, on the Meningitis B M14459 (fHbp) strain, one month after last vaccination; Test type: Other — M14459 strain- Between group ratio for comparison of MenABCWY group and rMenBOMV+ACWY_S group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 1.02, 80% CI 2-sided [0.86 to 1.22]
Statistical Analysis 10: Comparison: MenABCWY Group vs rMenBOMV+ACWY_S Group; Other unknown interference in MenABCWY versus rMenBOMV+ACWY_S study groups, on the Meningitis B 96217 (NadA)strain, one month after last vaccination; Test type: Other — 96217 strain- Between group ratio for comparison of MenABCWY group and rMenBOMV+ACWY_S group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.79, 80% CI 2-sided [0.66 to 0.95]
Statistical Analysis 11: Comparison: MenABCWY Group vs rMenBOMV+ACWY_S Group; Other unknown interference in MenABCWY versus rMenBOMV+ACWY_S study groups, on the Meningitis B NZ98/254 (PorA) strain, one month after last vaccination; Test type: Other — NZ98/254 strain- Between group ratio for comparison of MenABCWY group and rMenBOMV+ACWY_S group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.79, 80% CI 2-sided [0.65 to 0.97]
Statistical Analysis 12: Comparison: MenABCWY Group vs rMenBOMV+ACWY_S Group; Other unknown interference in MenABCWY versus rMenBOMV+ACWY_S study groups, on the Meningitis B M07-0241084 (NHBA) strain, one month after last vaccination; Test type: Non-Inferiority — M07-0241084 strain- Between group ratio for comparison of MenABCWY group and rMenBOMV+ACWY_S group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.73, 80% CI 2-sided [0.60 to 0.88]
Statistical Analysis 13: Comparison: MenABCWY Group vs rMenBOMV+ACWY_S Group; Other unknown interference in MenABCWY versus rMenBOMV+ACWY_S study groups, on the Meningitis serogrpoup A, one month after last vaccination; Test type: Other — Serogroup A- Between group ratio for comparison of MenABCWY group and rMenBOMV+ACWY_S group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.56, 80% CI 2-sided [0.45 to 0.69]
Statistical Analysis 14: Comparison: MenABCWY Group vs rMenBOMV+ACWY_S Group; Other unknown interference in MenABCWY versus rMenBOMV+ACWY_S study groups, on the Meningitis serogroup C, one month after last vaccination; Test type: Other — Serogroup C- Between group ratio for comparison of MenABCWY group and rMenBOMV+ACWY_S group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 1.19, 80% CI 2-sided [0.94 to 1.52]
Statistical Analysis 15: Comparison: MenABCWY Group vs rMenBOMV+ACWY_S Group; Other unknown interference in MenABCWY versus rMenBOMV+ACWY_S study groups, on the Meningitis serogroup W, one month after last vaccination; Test type: Other — Serogroup W- Between group ratio for comparison of MenABCWY group and rMenBOMV+ACWY_S group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 1.06, 80% CI 2-sided [0.87 to 1.29]
Statistical Analysis 16: Comparison: MenABCWY Group vs rMenBOMV+ACWY_S Group; Other unknown interference in MenABCWY versus rMenBOMV+ACWY_S study groups, on the Meningitis serogroup Y, one month after last vaccination; Test type: Other — Serogroup Y- Between group ratio for comparison of MenABCWY group and rMenBOMV+ACWY_S group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 1.18, 80% CI 2-sided [0.90 to 1.55]
Statistical Analysis 17: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_S versus rMenBOMV study groups, on the Meningitis B M14459(fHbp) strain, one month after last vaccination; Test type: Other — M14459 strain- Between group ratio for comparison of rMenBOMV+ACWY_S group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 1.02, 80% CI 2-sided [0.85 to 1.22]
Statistical Analysis 18: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_S versus rMenBOMV study groups, on the Meningitis B 96217 (NadA) strain, one month after last vaccination; Test type: Other — 96217 strain-Between group ratio for comparison of rMenBOMV+ACWY_S group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.90, 80% CI 2-sided [0.75 to 1.09]
Statistical Analysis 19: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_S versus rMenBOMV study groups, on the Meningitis B NZ98/254 (PorA) strain, one month after last vaccination; Test type: Other — NZ98/254 strain-Between group ratio for comparison of rMenBOMV+ACWY_S group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.78, 80% CI 2-sided [0.64 to 0.96]
Statistical Analysis 20: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_S versus rMenBOMV study groups, on the Meningitis B M07-0241084 (NHBA) strain, one month after last vaccination; Test type: Other — M07-0241084 strain-Between group ratio for comparison of rMenBOMV+ACWY_S group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.71, 80% CI 2-sided [0.58 to 0.86]
Statistical Analysis 21: Comparison: rMenBOMV+ACWY_S Group vs MenACWY Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_S versus MenACWY study groups, on the Meningitis serogroup A, one month after last vaccination; Test type: Other — Serogroup A- Between group ratio for comparison of rMenBOMV+ACWY_S group and MenACWY group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 3.60, 80% CI 2-sided [2.90 to 4.47]
Statistical Analysis 22: Comparison: rMenBOMV+ACWY_S Group vs MenACWY Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_S versus MenACWY study groups, on the Meningitis serogroup C, one month after last vaccination; Test type: Other — Serogroup C- Between group ratio for comparison of rMenBOMV+ACWY_S group and MenACWY group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 4.18, 80% CI 2-sided [3.28 to 5.31]
Statistical Analysis 23: Comparison: rMenBOMV+ACWY_S Group vs MenACWY Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_S versus MenACWY study groups, on the Meningitis serogroup W, one month after last vaccination; Test type: Other — Serogroup W- Between group ratio for comparison of rMenBOMV+ACWY_S group and MenACWY group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 3.07, 80% CI 2-sided [2.52 to 3.73]
Statistical Analysis 24: Comparison: rMenBOMV+ACWY_S Group vs MenACWY Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_S versus MenACWY study groups, on the Meningitis serogroup Y, one month after last vaccination; Test type: Other — Serogroup Y- Between group ratio for comparison of rMenBOMV+ACWY_S group and MenACWY group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 2.01, 80% CI 2-sided [1.53 to 2.65]
Statistical Analysis 25: Comparison: rMenBOMV+ACWY_D Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_D versus rMenBOMV study groups, on the Meningitis B M14459 (fHbp) strain, one month after last vaccination; Test type: Other — M14459 strain- Between group ratio for comparison of rMenBOMV+ACWY_D group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 1.02, 80% CI 2-sided [0.85 to 1.22]
Statistical Analysis 26: Comparison: rMenBOMV+ACWY_D Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_D versus rMenBOMV study groups, on the Meningitis B 96217 (NadA) strain, one month after last vaccination; Test type: Other — 96217 strain- Between group ratios for comparison of rMenBOMV+ACWY_D group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.86, 80% CI 2-sided [0.71 to 1.04]
Statistical Analysis 27: Comparison: rMenBOMV+ACWY_D Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_D versus rMenBOMV study groups, on the Meningitis B NZ98/254 (PorA) strain, one month after last vaccination; Test type: Other — NZ98/254 strain-Between group ratio for comparison of rMenBOMV+ACWY_D group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 1.01, 80% CI 2-sided [0.82 to 1.24]
Statistical Analysis 28: Comparison: rMenBOMV+ACWY_D Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_D versus rMenBOMV study groups, on the Meningitis B M07-0241084 (NHBA) strain, one month after last vaccination; Test type: Other — M07-0241084 strain-Between group ratio for comparison of rMenBOMV+ACWY_D group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.89, 80% CI 2-sided [0.73 to 1.09]
Statistical Analysis 29: Comparison: rMenBOMV+ACWY_D Group vs MenACWY Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_D versus MenACWY study groups, on the Meningitis serogroup A, one month after last vaccination; Test type: Other — Serogroup A-Between group ratio for comparison of rMenBOMV+ACWY_D group and MenACWY group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 3.92, 80% CI 2-sided [3.15 to 4.88]
Statistical Analysis 30: Comparison: rMenBOMV+ACWY_D Group vs MenACWY Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_D versus MenACWY study groups, on the Meningitis serogroup C, one month after last vaccination; Test type: Other — Serogroup C- Between group ratio for comparison of rMenBOMV+ACWY_D group and MenACWY group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 4.19, 80% CI 2-sided [3.30 to 5.34]
Statistical Analysis 31: Comparison: rMenBOMV+ACWY_D Group vs MenACWY Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_D versus MenACWY study groups, on the Meningitis serogroup W, one month after last vaccination; Test type: Other — Serogroup W- Between group ratio for comparison of rMenBOMV+ACWY_D group and MenACWY group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 3.17, 80% CI 2-sided [2.60 to 3.87]
Statistical Analysis 32: Comparison: rMenBOMV+ACWY_D Group vs MenACWY Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_D versus MenACWY study groups, on the Meningitis serogroup Y, one month after last vaccination; Test type: Other — Serogroup Y- Between group ratio for comparison of rMenBOMV+ACWY_D group and MenACWY group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 2.22, 80% CI 2-sided [1.68 to 2.92]
Statistical Analysis 33: Comparison: MenABCWY Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to MenABCWY versus rMenBOMV study groups, on the Meningitis B M14459 (fHbp) strain, one month after last vaccination; Test type: Other — M14459- Between group ratios for comparison of MenABCWY group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 1.05, 80% CI 2-sided [0.87 to 1.25]
Statistical Analysis 34: Comparison: MenABCWY Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to MenABCWY versus rMenBOMV study groups, on the Meningitis B 96217 (NadA) strain, one month after last vaccination; Test type: Other — 96217 strain- Between group ratio for comparison of MenABCWY group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.71, 80% CI 2-sided [0.59 to 0.86]
Statistical Analysis 35: Comparison: MenABCWY Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to MenABCWY versus rMenBOMV study groups, on the Meningitis B NZ98/254 (PorA) strain, one month after last vaccination; Test type: Other — NZ98/254 strain-Between group ratios for comparison of MenABCWY group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.62, 80% CI 2-sided [0.50 to 0.76]
Statistical Analysis 36: Comparison: MenABCWY Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to MenABCWY versus rMenBOMV study groups, on the Meningitis B M07-0241084 (NHBA) strain, one month after last vaccination; Test type: Other — M07-0241084 strain-Between group ratios for comparison of MenABCWY group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.52, 80% CI 2-sided [0.42 to 0.63]
Statistical Analysis 37: Comparison: MenABCWY Group vs MenACWY Group; To investigate possible effects on the immune response based on strains common to MenABCWY versus MenACWY study groups, on the Meningitis serogroup A, one month after last vaccination; Test type: Other — Serogroup A- Between group ratios for comparison between MenABCWY group and MenACWY group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 2.02, 80% CI 2-sided [1.62 to 2.51]
Statistical Analysis 38: Comparison: MenABCWY Group vs MenACWY Group; To investigate possible effects on the immune response based on strains common to MenABCWY versus MenACWY study groups, on the Meningitis serogroup C, one month after last vaccination; Test type: Other — Serogroup C- Between group ratios for comparison of MenABCWY group and MenACWY group; ANCOVA; The model is fitted to each serogroup/strain separately; Odds Ratio (OR) = 4.99, 80% CI 2-sided [3.92 to 6.35]
Statistical Analysis 39: Comparison: MenABCWY Group vs MenACWY Group; To investigate possible effects on the immune response based on strains common to MenABCWY versus MenACWY study groups, on the Meningitis serogroup W, one month after last vaccination; Test type: Other — Serogroup W- Between group ratios for comparison of MenABCWY group and MenACWY group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 3.25, 80% CI 2-sided [2.66 to 3.96]
Statistical Analysis 40: Comparison: MenABCWY Group vs MenACWY Group; To investigate possible effects on the immune response based on strains common to MenABCWY versus MenACWY study groups, on the Meningitis serogroup Y, one month after last vaccination; Test type: Other — Serogroup Y- Between group ratio for comparison of MenABCWY group and MenACWY group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 2.38, 80% CI 2-sided [1.81 to 3.12]

3. Primary Outcome: Percentage of Subjects With hSBA Titers Greater Than or Equal to(≥) the Lower Limit of Quantitation (LLOQ) Against Each of the N. Meningitidis Serogroup B Test Strains and Serogroups A, C, W-135 and Y,One Month After Last Vaccination.
Description: Immune responses against N. meningitidis serogroup B test strains and N. meningitidis serogroups A, C, W-135, and Y, were calculated in terms of percentage of subjects with hSBA titers ≥ LLOQ. Serogroup B strains tested were M14459 (factor H binding protein; fHbp), 96217 (Neisserial adhesin A; NadA), NZ98/254 (PorA), and M070241084 (Neisseria heparin binding antigen; NHBA).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (80% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY Group | rMenBOMV+ACWY_S Group | rMenBOMV+ACWY_D Group | rMenBOMV Group | MenACWY Group
Number analyzed (Participants) | 98 | 101 | 97 | 90 | 97
Percentage of subjects
  Meningitis B M14459 (fHbp): number analyzed (Participants) | 97 | 100 | 96 | 90 | 97
  Meningitis B M14459 (fHbp) | 83.5 [77.64 to 88.28] | 86.0 [80.50 to 90.35] | 88.5 [83.22 to 92.57] | 83.3 [77.18 to 88.31] | 12.4 [8.21 to 17.78]
  Mengitis B 96217(NadA): number analyzed (Participants) | 98 | 100 | 97 | 90 | 96
  Mengitis B 96217(NadA) | 96.9 [93.31 to 98.87] | 99.0 [96.17 to 99.89] | 99.0 [96.05 to 99.89] | 100.0 [97.47 to 100.00] | 33.3 [26.96 to 40.24]
  Meningitis B NZ98/254 (PorA): number analyzed (Participants) | 98 | 100 | 97 | 89 | 97
  Meningitis B NZ98/254 (PorA) | 59.2 [52.22 to 65.86] | 76.0 [69.66 to 81.53] | 80.4 [74.27 to 85.57] | 78.7 [72.05 to 84.23] | 5.2 [2.53 to 9.35]
  Meningitis B M07-0241084 (NHBA): number analyzed (Participants) | 98 | 100 | 96 | 89 | 95
  Meningitis B M07-0241084 (NHBA) | 59.2 [52.22 to 65.86] | 74.0 [67.54 to 79.71] | 77.1 [70.66 to 82.62] | 80.9 [74.48 to 86.22] | 23.2 [17.57 to 29.64]
  Meningitis A: number analyzed (Participants) | 97 | 101 | 97 | 90 | 93
  Meningitis A | 94.8 [90.65 to 97.47] | 100.0 [97.75 to 100.00] | 99.0 [96.05 to 99.89] | 91.1 [85.96 to 94.76] | 68.8 [61.86 to 75.15]
  Meningitis C: number analyzed (Participants) | 98 | 100 | 97 | 90 | 97
  Meningitis C | 100.0 [97.68 to 100.00] | 100.0 [97.72 to 100.00] | 100.0 [97.65 to 100.00] | 96.7 [92.73 to 98.77] | 86.6 [81.06 to 90.92]
  Meningitis W: number analyzed (Participants) | 98 | 100 | 96 | 90 | 97
  Meningitis W | 98.0 [94.66 to 99.46] | 96.0 [92.17 to 98.24] | 99.0 [96.01 to 99.89] | 93.3 [88.59 to 96.46] | 66.0 [59.09 to 72.36]
  Menngitis Y: number analyzed (Participants) | 97 | 100 | 97 | 89 | 96
  Menngitis Y | 99.0 [96.05 to 99.89] | 98.0 [94.77 to 99.47] | 96.9 [93.24 to 98.86] | 24.7 [18.79 to 31.54] | 85.4 [79.71 to 89.94]

4. Primary Outcome: Percentage of Subjects With a 4-fold Increase in hSBA Titers Against Each of the N. Meningitidis Serogroup B Test Strains and Against N. Meningitidis Serogroups A, C, W-135 and Y, One Month After Last Vaccination.
Description: Immune responses against N. meningitidis serogroup B test strains and N. meningitidis serogroups A, C, W-135, and Y, were calculated in terms of percentage of subjects with a 4-fold increase in hSBA titers. A 4-fold rise was defined as: a) for individuals whose pre-vaccination titers were less than (<) the limit of detection (LOD), the post-vaccination titers must have been ≥4-fold the LOD or ≥ the LLOQ, whichever was greater; b) for individuals whose pre-vaccination titers were ≥ the LOD and less than (<) the LLOQ, the post-vaccination titers must have been at least 4 times the LLOQ; and c) for individuals whose pre-vaccination titers were ≥ the LLOQ, the post-vaccination titers must have been at least 4 times the pre-vaccination titer. Serogroup B strains tested were M14459 (factor H binding protein; fHbp), 96217 (Neisserial adhesin A; NadA), NZ98/254 (PorA), and M070241084 (Neisseria heparin binding antigen; NHBA).
Time Frame: 1 month after last vaccination versus baseline (i.e.: at Day 91 versus Day 1 for all groups except the MenACWY Group, and at Day 31 versus Day 1 for the MenACWY Group).
Population: Analysis was performed on PPS for immunogenicity that included subjects who had no major protocol violations and whose assay results were available for at least 1 serogroup or B strain at Day 91 for all study groups except MenACWY Group or at Day 31 for the MenACWY Group and at baseline for all study groups.
Measure: Number (80% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY Group | rMenBOMV+ACWY_S Group | rMenBOMV+ACWY_D Group | rMenBOMV Group | MenACWY Group
Number analyzed (Participants) | 98 | 100 | 97 | 90 | 97
Percentage of subjects
  Meningitis B M14459 (fHbp): number analyzed (Participants) | 97 | 100 | 95 | 90 | 97
  Meningitis B M14459 (fHbp) | 66.0 [59.09 to 72.36] | 69.0 [62.32 to 75.09] | 66.3 [59.36 to 72.74] | 63.3 [56.09 to 70.11] | 2.1 [0.55 to 5.39]
  Meningitis B 96217(NadA): number analyzed (Participants) | 97 | 100 | 95 | 88 | 96
  Meningitis B 96217(NadA) | 80.4 [74.27 to 85.57] | 88.0 [82.74 to 92.04] | 90.5 [85.46 to 94.20] | 80.7 [74.20 to 86.06] | 2.1 [0.56 to 5.45]
  Meningitis B NZ98/254 (PorA): number analyzed (Participants) | 98 | 100 | 97 | 89 | 97
  Meningitis B NZ98/254 (PorA) | 48.0 [41.06 to 54.92] | 60.0 [53.11 to 66.58] | 58.8 [51.75 to 65.49] | 60.7 [53.35 to 67.63] | 1.0 [0.11 to 3.95]
  Meningitis B M07-0241084(NHBA): number analyzed (Participants) | 98 | 98 | 95 | 87 | 94
  Meningitis B M07-0241084(NHBA) | 21.4 [16.10 to 27.68] | 38.8 [32.18 to 45.72] | 42.1 [35.27 to 49.20] | 56.3 [48.88 to 63.54] | 2.1 [0.57 to 5.56]
  Meningitis A: number analyzed (Participants) | 96 | 100 | 95 | 90 | 92
  Meningitis A | 92.7 [88.04 to 95.90] | 99.0 [96.17 to 99.89] | 98.9 [95.97 to 99.89] | 87.8 [82.14 to 92.06] | 67.4 [60.34 to 73.85]
  Meningitis C: number analyzed (Participants) | 98 | 99 | 97 | 89 | 96
  Meningitis C | 90.8 [85.89 to 94.38] | 91.9 [87.21 to 95.24] | 86.6 [81.06 to 90.92] | 57.3 [49.95 to 64.40] | 52.1 [45.05 to 59.05]
  Meningitis W: number analyzed (Participants) | 96 | 98 | 93 | 85 | 95
  Meningitis W | 83.3 [77.41 to 88.15] | 78.6 [72.32 to 83.90] | 74.2 [67.48 to 80.10] | 74.1 [67.04 to 80.30] | 41.1 [34.26 to 48.14]
  Meningitis Y: number analyzed (Participants) | 97 | 99 | 95 | 88 | 95
  Meningitis Y | 95.9 [91.93 to 98.19] | 91.9 [87.21 to 95.24] | 93.7 [89.18 to 96.65] | 11.4 [7.19 to 16.97] | 76.8 [70.36 to 82.43]

5. Primary Outcome: hSBA Adjusted Geometric Mean Ratios (GMRs) Against Each of the N. Meningitidis Serogroup B Test Strains and Against N. Meningitidis Serogroups A, C, W-135 and Y, One Month After Last Vaccination.
Description: hSBA mean ratios at 1 month after the last vaccination versus baseline were calculated in terms of GMRs i.e. as the anti-logarithm of the mean of the change from baseline of log-transformed titer values at 1 month after last vaccination and Baseline. Serogroup B strains tested were M14459 (factor H binding protein; fHbp), 96217 (Neisserial adhesin A; NadA), NZ98/254 (PorA), and M070241084 (Neisseria heparin binding antigen; NHBA). Adjusted means were obtained from ANCOVA model fitted to each Serogroup (Strain) individually, study group and center as fixed effects and zero-centered pre-vaccination log-transformed titer as a continuous covariate.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (80% Confidence Interval); unit: Ratio
Arm/Group | MenABCWY Group | rMenBOMV+ACWY_S Group | rMenBOMV+ACWY_D Group | rMenBOMV Group | MenACWY Group
Number analyzed (Participants) | 98 | 100 | 97 | 90 | 97
Ratio
  Meningitis B M14459 (fHbp): number analyzed (Participants) | 97 | 100 | 95 | 90 | 97
  Meningitis B M14459 (fHbp) | 11.17 [9.59 to 13.02] | 10.90 [9.42 to 12.62] | 10.85 [9.30 to 12.66] | 10.69 [9.12 to 12.52] | 1.16 [0.99 to 1.35]
  Meningitis B 96217(NadA): number analyzed (Participants) | 97 | 100 | 95 | 88 | 96
  Meningitis B 96217(NadA) | 21.33 [18.22 to 24.99] | 27.02 [23.22 to 31.44] | 25.66 [21.88 to 30.10] | 29.87 [25.32 to 35.24] | 1.09 [0.93 to 1.28]
  Meningitis B NZ98/254(PorA): number analyzed (Participants) | 98 | 100 | 97 | 89 | 97
  Meningitis B NZ98/254(PorA) | 7.28 [6.11 to 8.67] | 9.20 [7.78 to 10.88] | 11.85 [9.94 to 14.13] | 11.77 [9.81 to 14.12] | 1.21 [1.01 to 1.44]
  Meningitis B M07-0241084(NHBA): number analyzed (Participants) | 98 | 98 | 95 | 87 | 94
  Meningitis B M07-0241084(NHBA) | 3.60 [3.05 to 4.25] | 4.96 [4.23 to 5.81] | 6.22 [5.27 to 7.35] | 6.98 [5.87 to 8.30] | 1.12 [0.95 to 1.33]
  Meningitis A: number analyzed (Participants) | 96 | 100 | 95 | 90 | 92
  Meningitis A | 33.21 [27.55 to 40.04] | 59.36 [49.68 to 70.93] | 64.58 [53.52 to 77.93] | 30.05 [24.77 to 36.44] | 16.47 [13.62 to 19.93]
  Meningitis C: number analyzed (Participants) | 98 | 99 | 97 | 89 | 96
  Meningitis C | 34.34 [27.88 to 42.30] | 28.74 [23.52 to 35.13] | 28.86 [23.40 to 35.60] | 6.35 [5.11 to 7.90] | 6.88 [5.58 to 8.49]
  Meningitis W: number analyzed (Participants) | 96 | 98 | 93 | 85 | 95
  Meningitis W | 24.58 [20.72 to 29.15] | 23.21 [19.69 to 27.36] | 24.02 [20.20 to 28.56] | 18.29 [15.28 to 21.90] | 7.57 [6.37 to 8.99]
  Meningitis Y: number analyzed (Participants) | 97 | 99 | 95 | 88 | 95
  Meningitis Y | 106.87 [84.27 to 135.53] | 90.59 [72.18 to 113.70] | 99.76 [78.58 to 126.66] | 1.78 [1.39 to 2.28] | 44.99 [35.42 to 57.14]

6. Secondary Outcome: hSBA Adjusted GMTs Against All of N. Meningitidis Serogroup B Test Strains (Pooled), One Month After First Vaccination
Description: as for outcome 1
Time Frame: 1 month after first vaccination i.e.: at Day 31 for all groups except for the MenACWY Group
Population: Analysis was performed on PPS for immunogenicity that included subjects who had no major protocol violations and whose assay results were available for at least 1 serogroup or B strain after first vaccination for all study groups except for MenACWY group that was not considered for this analysis as only serogroup B strains assessed in this outcome.
Measure: Geometric Mean (80% Confidence Interval); unit: Titers
Arm/Group | MenABCWY Group | rMenBOMV+ACWY_S Group | rMenBOMV+ACWY_D Group | rMenBOMV Group
Number analyzed (Participants) | 96 | 103 | 98 | 91
Titers | 6.51 [5.63 to 7.52] | 8.33 [7.24 to 9.58] | 8.16 [7.08 to 9.41] | 9.45 [8.14 to 10.95]
Statistical Analysis 1: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV+ACWY_D Group; Immune interference due to stress to lymph nodes (lymph-node effect) in rMenBOMV+ACWY_S versus rMenBOMV+ACWY_D study groups, on the pooled B strains, one month after first vaccination; Test type: Other — Between group ratio is calculated as GMT for rMenBOMV+ACWY_S Group over GMT for rMenBOMV+ACWY_D Group. 80% CI are obtained from Analysis of Covariance model fitted to pooled Serogroup B Strains. The following ANCOVA model is used: fixed-effect model including age strata, study group, strain and center as fixed effects. The pre vaccination (Baseline) log-transformed titer with centering at zero is included as a continuous covariate; ANCOVA; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio = 1.02, 80% CI 2-sided [0.86 to 1.22]

7. Secondary Outcome: hSBA Adjusted GMTs Against Each of the N. Meningitidis Serogroup B Test Strains and N. Meningitidis Serogroups A, C, W-135 and Y, One Month After First Vaccination.
Description: as for outcome 2
Time Frame: 1 month after first vaccination i.e.: at Day 31 for all groups except for the MenACWY Group.
Population: Analysis was performed on PPS for immunogenicity that included subjects who had no major protocol violations and whose assay results were available for at least 1 serogroup/ B strain after first vaccination for all study groups except for MenACWY Group for which results were included in the last vaccination analysis (see primary outcome measure 2).
Measure: Geometric Mean (80% Confidence Interval); unit: Titers
Arm/Group | MenABCWY Group | rMenBOMV+ACWY_S Group | rMenBOMV+ACWY_D Group | rMenBOMV Group
Number analyzed (Participants) | 96 | 103 | 98 | 91
Titers
  Meningitis B M14459(fHbp): number analyzed (Participants) | 95 | 103 | 98 | 90
  Meningitis B M14459(fHbp) | 5.50 [4.55 to 6.66] | 6.36 [5.29 to 7.65] | 4.94 [4.09 to 5.96] | 6.08 [5.00 to 7.39]
  Meningitis B 96217 (NadA) | 8.21 [6.87 to 9.81] | 11.30 [9.51 to 13.42] | 12.18 [10.23 to 14.52] | 14.07 [11.72 to 16.89]
  Meningitis B NZ98/254 (PorA): number analyzed (Participants) | 96 | 103 | 98 | 90
  Meningitis B NZ98/254 (PorA) | 3.79 [3.10 to 4.63] | 4.83 [3.98 to 5.86] | 4.76 [3.91 to 5.79] | 5.48 [4.47 to 6.71]
  Meningitis B M07-0241084 (NHBA): number analyzed (Participants) | 94 | 101 | 96 | 90
  Meningitis B M07-0241084 (NHBA) | 6.27 [5.23 to 7.52] | 7.31 [6.12 to 8.73] | 6.75 [5.65 to 8.06] | 7.69 [6.38 to 9.26]
  Meningitis A: number analyzed (Participants) | 95 | 102 | 96 | 90
  Meningitis A | 31.38 [24.79 to 39.73] | 67.95 [54.07 to 85.40] | 88.29 [69.95 to 111.44] | 8.22 [6.48 to 10.44]
  Meningitis C: number analyzed (Participants) | 96 | 102 | 97 | 90
  Meningitis C | 41.35 [32.39 to 52.79] | 33.76 [26.61 to 42.85] | 40.33 [31.71 to 51.29] | 11.47 [8.92 to 14.74]
  Meningitis W: number analyzed (Participants) | 96 | 102 | 97 | 88
  Meningitis W | 108.91 [88.67 to 133.78] | 81.38 [66.62 to 99.42] | 92.84 [75.75 to 113.80] | 42.99 [34.66 to 53.33]
  Meningitis Y: number analyzed (Participants) | 95 | 99 | 95 | 90
  Meningitis Y | 75.07 [56.86 to 99.13] | 76.48 [58.31 to 100.32] | 100.30 [76.13 to 132.15] | 3.98 [3.00 to 5.30]
Statistical Analysis 1: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV+ACWY_D Group; Immune interference due to stress to lymph nodes (lymph-node effect) in rMenBOMV+ACWY_S versus rMenBOMV+ACWY_D study groups, on the Meningitis B M14459 (fHbp) strain, one month after first vaccination; Test type: Other — M14459 strain- Between group ratio for comparison of rMenBOMV+ACWY_S group and rMenBOMV+ACWY_D group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 1.29, 80% CI 2-sided [1.02 to 1.63]
Statistical Analysis 2: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV+ACWY_D Group; Immune interference due to stress to lymph nodes (lymph-node effect) in rMenBOMV+ACWY_S versus rMenBOMV+ACWY_D study groups, on the Meningitis B 96217 (NadA) strain, one month after first vaccination; Test type: Other — 96217 strain- Between group ratio for comparison of rMenBOMV+ACWY_S group and rMenBOMV+ACWY_D group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.93, 80% CI 2-sided [0.75 to 1.15]
Statistical Analysis 3: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV+ACWY_D Group; Immune interference due to stress to lymph nodes (lymph-node effect) in rMenBOMV+ACWY_S versus rMenBOMV+ACWY_D study groups, on the Meningitis B NZ98/254 (PorA)strain, one month after first vaccination; Test type: Other — NZ98/254 strain- Between group ratio for comparison of rMenBOMV+ACWY_S group and rMenBOMV+ACWY_D group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 1.01, 80% CI 2-sided [0.80 to 1.29]
Statistical Analysis 4: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV+ACWY_D Group; Immune interference due to stress to lymph nodes (lymph-node effect) in rMenBOMV+ACWY_S versus rMenBOMV+ACWY_D study groups, on the Meningitis B M07-0241084 (NHBA) strain, one month after first vaccination; Test type: Other — M07-0241084 strain-Between group ratio for comparison of rMenBOMV+ACWY_S group and rMenBOMV+ACWY_D group; ANCOVA; The model is fitted to each serogroup/strain separately; Odds Ratio (OR) = 1.08, 80% CI 2-sided [0.87 to 1.36]
Statistical Analysis 5: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV+ACWY_D Group; Immune interference due to stress to lymph nodes (lymph-node effect) in rMenBOMV+ACWY_S versus rMenBOMV+ACWY_D study groups, on the Meningitis serogroup A, one month after first vaccination; Test type: Other — Serogroup A- Between group ratio for comparison of rMenBOMV+ACWY_S group and rMenBOMV+ACWY_D group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.77, 80% CI 2-sided [0.58 to 1.03]
Statistical Analysis 6: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV+ACWY_D Group; Immune interference due to stress to lymph nodes (lymph-node effect) in rMenBOMV+ACWY_S versus rMenBOMV+ACWY_D study groups, on the Meningitis serogroup C, one month after first vaccination; Test type: Other — Serogroup C- Between group ratio for comparison of rMenBOMV+ACWY_S group and rMenBOMV+ACWY_D Group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.84, 80% CI 2-sided [0.62 to 1.13]
Statistical Analysis 7: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV+ACWY_D Group; Immune interference due to stress to lymph nodes (lymph-node effect) in rMenBOMV+ACWY_S versus rMenBOMV+ACWY_D study groups, on the Meningitis serogroup W, one month after first vaccination; Test type: Other — Serogroup W- Between group ratio for comparison of rMenBOMV+ACWY_S group and rMenBOMV+ACWY_D group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.88, 80% CI 2-sided [0.68 to 1.13]
Statistical Analysis 8: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV+ACWY_D Group; Immune interference due to stress to lymph nodes (lymph-node effect) in rMenBOMV+ACWY_S versus rMenBOMV+ACWY_D study groups, on the Meningitis serogroup Y, one month after first vaccination; Test type: Other — Serogroup Y- Between group ratio for comparison of rMenBOMV+ACWY_S group and rMenBOMV+ACWY_D group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.76, 80% CI 2-sided [0.54 to 1.08]
Statistical Analysis 9: Comparison: MenABCWY Group vs rMenBOMV+ACWY_S Group; Other unknown interference in MenABCWY versus rMenBOMV+ACWY_S study groups, on the Meningitis B M14459 (fHbp) strain, one month after first vaccination; Test type: Other — M14459 strain- Between group ratio for comparison of MenABCWY group and rMenBOMV+ACWY_S group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.87, 80% CI 2-sided [0.69 to 1.09]
Statistical Analysis 10: Comparison: MenABCWY Group vs rMenBOMV+ACWY_S Group; Other unknown interference in MenABCWY versus rMenBOMV+ACWY_S study groups, on the Meningitis B 96217 (NadA) strain, one month after first vaccination; Test type: Other — 96217 strain- Between group ratio for comparison of MenABCWY group and rMenBOMV+ACWY_S group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.73, 80% CI 2-sided [0.58 to 0.90]
Statistical Analysis 11: Comparison: MenABCWY Group vs rMenBOMV+ACWY_S Group; Other unknown interference in MenABCWY versus rMenBOMV+ACWY_S study groups, on the Meningitis B NZ98/254 (PorA) strain, one month after first vaccination; Test type: Other — NZ98/254 strain- Between group ratio for comparison of MenABCWY group and rMenBOMV+ACWY_S group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.78, 80% CI 2-sided [0.61 to 1.00]
Statistical Analysis 12: Comparison: MenABCWY Group vs rMenBOMV+ACWY_S Group; Other unknown interference in MenABCWY versus rMenBOMV+ACWY_S study groups, on the Meningitis B M07-0241084 (NHBA) strain, one month after first vaccination; Test type: Other — M07-0241084 strain- Between group ratio for comparison of MenABCWY group and rMenBOMV+ACWY_S group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.86, 80% CI 2-sided [0.68 to 1.07]
Statistical Analysis 13: Comparison: MenABCWY Group vs rMenBOMV+ACWY_S Group; Other unknown interference in MenABCWY versus rMenBOMV+ACWY_S study groups, on the Meningitis serogroup A, one month after first vaccination; Test type: Other — Serogroup A- Between group ratio for comparison of MenABCWY group and rMenBOMV+ACWY_S group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.46, 80% CI 2-sided [0.35 to 0.62]
Statistical Analysis 14: Comparison: MenABCWY Group vs rMenBOMV+ACWY_S Group; Other unknown interference in MenABCWY versus rMenBOMV+ACWY_S study groups, on the Meningitis serogroup C, one month after first vaccination; Test type: Other — Serogroup C- Between group ratio for comparison of MenABCWY group and rMenBOMV+ACWY_S group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 1.22, 80% CI 2-sided [0.91 to 1.65]
Statistical Analysis 15: Comparison: MenABCWY Group vs rMenBOMV+ACWY_S Group; Other unknown interference in MenABCWY versus rMenBOMV+ACWY_S study groups, on the Meningitis serogroup W, one month after first vaccination; Test type: Other — Serogroup W- Between group ratio for comparison of MenABCWY group and rMenBOMV+ACWY_S group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 1.34, 80% CI 2-sided [1.04 to 1.72]
Statistical Analysis 16: Comparison: MenABCWY Group vs rMenBOMV+ACWY_S Group; Other unknown interference in MenABCWY versus rMenBOMV+ACWY_S study groups, on the Meningitis serogroup Y, one month after first vaccination; Test type: Other — Serogroup Y- Between group ratio for comparison of MenABCWY group and rMenBOMV+ACWY_S group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.98, 80% CI 2-sided [0.70 to 1.38]
Statistical Analysis 17: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_S versus rMenBOMV study groups, on the Meningitis B M14459 (fHbp) strain, one month after first vaccination; Test type: Other — M14459 strain-Between group ratio for comparison of rMenBOMV_ACWY_S group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 1.05, 80% CI 2-sided [0.83 to 1.32]
Statistical Analysis 18: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_S versus rMenBOMV study groups, on the Meningitis B 96217 (NadA) strain, one month after first vaccination; Test type: Other — 96217 strain-Between group ratio for comparison of rMenBOMV_ACWY_S group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.80, 80% CI 2-sided [0.64 to 1.00]
Statistical Analysis 19: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_S versus rMenBOMV study groups, on the Meningitis B NZ98/254 (PorA) strain, one month after first vaccination; Test type: Other — NZ98/254 strain -Between group ratio for comparison of rMenBOMV_ACWY_S group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.88, 80% CI 2-sided [0.69 to 1.13]
Statistical Analysis 20: Comparison: rMenBOMV+ACWY_S Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_S versus rMenBOMV study groups, on the Meningitis B M07-0241084 (NHBA) strain, one month after first vaccination; Test type: Other — M07-0241084 strain -Between group ratio for comparison of rMenBOMV_ACWY_S group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.95, 80% CI 2-sided [0.76 to 1.19]
Statistical Analysis 21: Comparison: rMenBOMV+ACWY_D Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_D versus rMenBOMV study groups, on the Meningitis B M14459 (fHbp) strain, one month after first vaccination; Test type: Other — M14459 strain -Between group ratio for comparison of rMenBOMV_ACWY_D group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.81, 80% CI 2-sided [0.64 to 1.03]
Statistical Analysis 22: Comparison: rMenBOMV+ACWY_D Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_D versus rMenBOMV study groups, on the Meningitis B 96217 (NadA) strain, one month after first vaccination; Test type: Other — 96217 strain -Between group ratio for comparison of rMenBOMV_ACWY_D group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.87, 80% CI 2-sided [0.69 to 1.09]
Statistical Analysis 23: Comparison: rMenBOMV+ACWY_D Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_D versus rMenBOMV study groups, on the Meningitis B NZ98/254 (PorA) strain, one month after first vaccination; Test type: Other — NZ98/254 strain -Between group ratio for comparison of rMenBOMV_ACWY_D group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometrical mean ratio = 0.87, 80% CI 2-sided [0.68 to 1.12]
Statistical Analysis 24: Comparison: rMenBOMV+ACWY_D Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to rMenBOMV+ACWY_D versus rMenBOMV study groups, on the Meningitis B M07-0241084 (NHBA) strain, one month after first vaccination; Test type: Other — M07-0241084 strain-Between group ratio for comparison of rMenBOMV_ACWY_D group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometrical mean ratio = 0.88, 80% CI 2-sided [0.70 to 1.10]
Statistical Analysis 25: Comparison: MenABCWY Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to MenABCWY versus rMenBOMV study groups, on the Meningitis B M14459 (fHbp)strain, one month after first vaccination; Test type: Other — M14459 strain-Between group ratio for comparison of MenABCWY group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.91, 80% CI 2-sided [0.71 to 1.15]
Statistical Analysis 26: Comparison: MenABCWY Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to MenABCWY versus rMenBOMV study groups, on the Meningitis B 96217 (NadA) strain, one month after first vaccination; Test type: Other — 96217 strain-Between group ratio for comparison of MenABCWY group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.58, 80% CI 2-sided [0.47 to 0.73]
Statistical Analysis 27: Comparison: MenABCWY Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to MenABCWY versus rMenBOMV study groups, on the Meningitis B NZ98/254 (PorA) strain, one month after first vaccination; Test type: Other — NZ98/254 strain-Between group ratio for comparison of MenABCWY group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.69, 80% CI 2-sided [0.54 to 0.89]
Statistical Analysis 28: Comparison: MenABCWY Group vs rMenBOMV Group; To investigate possible effects on the immune response based on strains common to MenABCWY versus rMenBOMV study groups, on the Meningitis B M07-0241084 (NHBA) strain, one month after first vaccination; Test type: Other — M07-0241084 strain-Between group ratio for comparison of MenABCWY group and rMenBOMV group; ANCOVA; The model is fitted to each serogroup/strain separately; Geometric mean ratio = 0.82, 80% CI 2-sided [0.65 to 1.03]

8. Secondary Outcome: Percentage of Subjects With hSBA Titers Greater Than or Equal to (≥) the LLOQ Against Each of the N. Meningitidis Serogroup B Test Strains and Against Serogroups A, C, W-135, and Y, One Month After First Vaccination
Description: as for outcome 3
Time Frame: 1 month after first vaccination i.e.: at Day 31 for all groups except for the MenACWY Group
Population: Analysis was performed on PPS for immunogenicity that included subjects who had no major protocol violations and whose assay results were available for at least 1 serogroup/B strain after first vaccination for all study groups except for MenACWY Group for which results were included in the last vaccination analysis (see primary outcome measure 3).
Measure: Number (80% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY Group | rMenBOMV+ACWY_S Group | rMenBOMV+ACWY_D Group | rMenBOMV Group
Number analyzed (Participants) | 96 | 103 | 98 | 91
Percentage of subjects
  Meningitis B M14459 (fHbp): number analyzed (Participants) | 95 | 103 | 98 | 90
  Meningitis B M14459 (fHbp) | 36.8 [30.24 to 43.88] | 49.5 [42.77 to 56.27] | 37.8 [31.21 to 44.69] | 42.2 [35.19 to 49.53]
  Meningitis B 96217 (NadA) | 57.3 [50.24 to 64.11] | 66.0 [59.35 to 72.20] | 69.4 [62.65 to 75.51] | 75.8 [69.12 to 81.64]
  Meningitis B NZ98/254 (PorA): number analyzed (Participants) | 96 | 103 | 98 | 90
  Meningitis B NZ98/254 (PorA) | 29.2 [23.08 to 35.93] | 37.9 [31.48 to 44.61] | 33.7 [27.35 to 40.51] | 37.8 [30.94 to 45.04]
  Meningitis B M07-0241084 (NHBA): number analyzed (Participants) | 94 | 101 | 96 | 90
  Meningitis B M07-0241084 (NHBA) | 35.1 [28.56 to 42.14] | 49.5 [42.69 to 56.33] | 37.5 [30.90 to 44.51] | 44.4 [37.33 to 51.75]
  Meningitis A: number analyzed (Participants) | 95 | 102 | 96 | 90
  Meningitis A | 65.3 [58.28 to 71.75] | 73.5 [67.12 to 79.22] | 80.2 [74.01 to 85.41] | 25.6 [19.58 to 32.38]
  Meningitis C: number analyzed (Participants) | 96 | 102 | 97 | 90
  Meningitis C | 89.6 [84.41 to 93.42] | 94.1 [89.90 to 96.88] | 92.8 [88.16 to 95.94] | 70.0 [62.96 to 76.35]
  Meningitis W: number analyzed (Participants) | 96 | 102 | 97 | 88
  Meningitis W | 71.9 [65.16 to 77.88] | 70.6 [64.04 to 76.51] | 74.2 [67.67 to 80.00] | 52.3 [44.90 to 59.56]
  Meningitis Y: number analyzed (Participants) | 95 | 99 | 95 | 90
  Meningitis Y | 83.2 [77.18 to 88.02] | 81.8 [75.86 to 86.76] | 88.4 [83.05 to 92.49] | 20.0 [14.60 to 26.45]

9. Secondary Outcome: Percentage of Subjects With a 4-fold Increase in hSBA Titers Against Each of the N. Meningitidis Serogroup B Test Strains and Against N. Meningitidis Serogroups A, C, W-135, and Y, One Month After First Vaccination
Description: Immune responses against N. meningitidis serogroup B test strains and N. meningitidis serogroups A, C, W-135, and Y, were calculated in terms of percentage of subjects with a 4-fold increase in hSBA titers. A 4-fold rise is defined as: a) for individuals whose pre-vaccination titers were less than (<) the limit of detection (LOD), the post-vaccination titers must have been ≥4-fold the LOD or ≥ the LLOQ, whichever was greater; b) for individuals whose pre-vaccination titers were ≥ the LOD and less than (<) the LLOQ, the post-vaccination titers must have been at least 4 times the LLOQ; and c) for individuals whose pre-vaccination titers were ≥ the LLOQ, the post-vaccination titers must have been at least 4 times the pre-vaccination titer. Serogroup B strains tested were M14459 (factor H binding protein; fHbp), 96217 (Neisserial adhesin A; NadA), NZ98/254 (PorA), and M070241084 (Neisseria heparin binding antigen; NHBA).
Time Frame: 1 month after first vaccination versus baseline (i.e.: at Day 31 versus Day 1 for all groups except for the MenACWY Group)
Population: Analysis was performed on PPS for immunogenicity that included subjects who had no major protocol violations and whose assay results were available for at least 1 serogroup/B strain after first vaccination for all study groups except for MenACWY Group for which results were included in the last vaccination analysis (see primary outcome measure 4).
Measure: Number (80% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY Group | rMenBOMV+ACWY_S Group | rMenBOMV+ACWY_D Group | rMenBOMV Group
Number analyzed (Participants) | 96 | 103 | 97 | 91
Percentage of subjects
  Meningitis B M14459 (fHbp): number analyzed (Participants) | 95 | 103 | 96 | 90
  Meningitis B M14459 (fHbp) | 24.2 [18.52 to 30.76] | 24.3 [18.80 to 30.53] | 18.8 [13.67 to 24.86] | 25.6 [19.58 to 32.38]
  Meningitis B 96217 (NadA): number analyzed (Participants) | 95 | 103 | 95 | 89
  Meningitis B 96217 (NadA) | 22.1 [16.62 to 28.51] | 34.0 [27.80 to 40.65] | 30.5 [24.31 to 37.38] | 32.6 [26.01 to 39.77]
  Meningitis B NZ98/254 (PorA): number analyzed (Participants) | 96 | 103 | 97 | 90
  Meningitis B NZ98/254 (PorA) | 20.8 [15.51 to 27.11] | 26.2 [20.57 to 32.58] | 26.8 [20.94 to 33.42] | 27.8 [21.60 to 34.72]
  Meningitis B M07-0241084 (NHBA): number analyzed (Participants) | 94 | 97 | 94 | 88
  Meningitis B M07-0241084 (NHBA) | 9.6 [5.86 to 14.69] | 20.6 [15.35 to 26.84] | 13.8 [9.37 to 19.52] | 20.5 [14.94 to 27.03]
  Meningitis A: number analyzed (Participants) | 94 | 101 | 93 | 90
  Meningitis A | 61.7 [54.60 to 68.42] | 71.3 [64.73 to 77.18] | 80.6 [74.37 to 85.88] | 23.3 [17.57 to 30.03]
  Meningitis C: number analyzed (Participants) | 96 | 101 | 96 | 89
  Meningitis C | 54.2 [47.11 to 61.09] | 46.5 [39.78 to 53.39] | 51.0 [44.02 to 58.03] | 24.7 [18.79 to 31.54]
  Meningitis W: number analyzed (Participants) | 94 | 100 | 93 | 83
  Meningitis W | 60.6 [53.53 to 67.40] | 52.0 [45.12 to 58.82] | 51.6 [44.46 to 58.71] | 39.8 [32.53 to 47.37]
  Meningitis Y: number analyzed (Participants) | 95 | 98 | 92 | 89
  Meningitis Y | 77.9 [71.49 to 83.38] | 75.5 [69.06 to 81.14] | 78.3 [71.76 to 83.79] | 9.0 [5.30 to 14.19]

10. Secondary Outcome: hSBA Adjusted GMRs Against Each of the N. Meningitidis Serogroup B Test Strains and Against N. Meningitidis Serogroups A, C, W-135, and Y, One Month After First Vaccination
Description: hSBA mean ratios at 1 month after the first vaccination versus baseline were calculated in terms of GMRs. i.e. as the anti-logarithm of the mean of the change from baseline of log-transformed titer values at 1 month after first vaccination and Baseline. Serogroup B strains tested were M14459 (factor H binding protein; fHbp), 96217 (Neisserial adhesin A; NadA), NZ98/254 (PorA), and M070241084 (Neisseria heparin binding antigen; NHBA). Adjusted mean were obtained from ANCOVA model fitted to each Serogroup (Strain) individually, study group and center as fixed effects and zero-centered pre-vaccination log-transformed titer as a continuous covariate.
Time Frame: as for outcome 9
Population: Analysis was performed on PPS for immunogenicity that included subjects who had no major protocol violations and whose assay results were available for at least 1 serogroup/B strain after first vaccination for all study groups except for MenACWY Group for which results were included in the last vaccination analysis (see primary outcome measure 5).
Measure: Geometric Mean (80% Confidence Interval); unit: Ratio
Arm/Group | MenABCWY Group | rMenBOMV+ACWY_S Group | rMenBOMV+ACWY_D Group | rMenBOMV Group
Number analyzed (Participants) | 96 | 103 | 97 | 90
Ratio
  Meningitis B M14459 (fHbp): number analyzed (Participants) | 95 | 103 | 96 | 90
  Meningitis B M14459 (fHbp) | 2.59 [2.14 to 3.14] | 3.00 [2.49 to 3.61] | 2.33 [1.93 to 2.81] | 2.87 [2.36 to 3.48]
  Meningitis B 96217(NadA): number analyzed (Participants) | 95 | 103 | 95 | 89
  Meningitis B 96217(NadA) | 2.15 [1.80 to 2.57] | 2.96 [2.49 to 3.51] | 3.19 [2.68 to 3.80] | 3.68 [3.07 to 4.42]
  Meningitis B NZ98/254 (PorA) | 2.16 [1.77 to 2.64] | 2.76 [2.27 to 3.34] | 2.72 [2.23 to 3.31] | 3.13 [2.55 to 3.83]
  Meningitis B M07-0241084 (NHBA): number analyzed (Participants) | 94 | 97 | 94 | 88
  Meningitis B M07-0241084 (NHBA) | 1.73 [1.44 to 2.07] | 2.01 [1.69 to 2.41] | 1.86 [1.56 to 2.22] | 2.12 [1.76 to 2.55]
  Meningitis A: number analyzed (Participants) | 94 | 101 | 93 | 90
  Meningitis A | 10.15 [8.02 to 12.85] | 21.97 [17.48 to 27.62] | 28.55 [22.62 to 36.04] | 2.66 [2.09 to 3.38]
  Meningitis C: number analyzed (Participants) | 96 | 101 | 96 | 89
  Meningitis C | 8.08 [6.33 to 10.31] | 6.59 [5.20 to 8.37] | 7.88 [6.19 to 10.02] | 2.24 [1.74 to 2.88]
  Meningitis W: number analyzed (Participants) | 94 | 100 | 93 | 83
  Meningitis W | 11.08 [9.02 to 13.60] | 8.28 [6.77 to 10.11] | 9.44 [7.70 to 11.57] | 4.37 [3.52 to 5.42]
  Meningitis Y: number analyzed (Participants) | 95 | 98 | 92 | 89
  Meningitis Y | 36.58 [27.70 to 48.30] | 37.26 [28.41 to 48.88] | 48.87 [37.09 to 64.39] | 1.94 [1.46 to 2.58]

11. Secondary Outcome: Number of Subjects With Any Solicited Local Adverse Events (AEs)
Description: Assessed local AEs were erythema, swelling, induration and pain. Any erythema, swelling and induration is defined as a symptom with a surface diameter equal to or greater than 25 millimeters.
Time Frame: During the 7 days (including the day of vaccination) after each vaccination i.e after Dose 1 administered at Day 1 (for all groups) and after Dose 2 administered at Day 61 (for all groups except for MenACWY Group)
Population: Analysis was performed on solicited safety set that included all subjects who provided informed consent,underwent screening procedures,had a subject number assigned,received a study vaccination & was reported with any solicited adverse event data.No results for dose 2 categories for subjects of MenACWY Group as they received only 1 dose at day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | MenABCWY Group | rMenBOMV+ACWY_S Group | rMenBOMV+ACWY_D Group | rMenBOMV Group | MenACWY Group
Number analyzed (Participants) | 100 | 104 | 100 | 94 | 102
Participants
  Erythema at Dose 1 | 17 | 19 | 18 | 9 | 7
  Swelling at Dose 1 | 20 | 21 | 16 | 13 | 10
  Induration at Dose 1 | 9 | 15 | 12 | 6 | 4
  Pain at Dose 1 | 89 | 100 | 95 | 88 | 52
  Erythema at Dose 2: number analyzed (Participants) | 100 | 104 | 100 | 94 | 0
  Erythema at Dose 2 | 15 | 18 | 15 | 10 |
  Swelling at Dose 2: number analyzed (Participants) | 100 | 104 | 100 | 94 | 0
  Swelling at Dose 2 | 13 | 14 | 15 | 12 |
  Induration at Dose 2: number analyzed (Participants) | 100 | 104 | 100 | 94 | 0
  Induration at Dose 2 | 6 | 11 | 12 | 12 |
  Pain at Dose 2: number analyzed (Participants) | 100 | 104 | 100 | 94 | 0
  Pain at Dose 2 | 87 | 97 | 95 | 87 |

12. Secondary Outcome: Number of Subjects With Any Solicited Systemic AEs
Description: Assessed systemic AEs were arthralgia, fatigue, nausea, headache, myalgia and fever. Any fever is defined as body temperature equal or greater than 38 degrees Celsius.
Time Frame: as for outcome 11
Population: Analysis was performed on solicited safety set that included all subjects who provided informed consent,underwent screening procedures,had a subject number assigned,received a study vaccination & was reported with any solicited adverse event data.No results for dose 2 category for subjects of MenACWY Group as they received only 1 dose at day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | MenABCWY Group | rMenBOMV+ACWY_S Group | rMenBOMV+ACWY_D Group | rMenBOMV Group | MenACWY Group
Number analyzed (Participants) | 100 | 104 | 100 | 94 | 102
Participants
  Arthralgia at Dose 1: number analyzed (Participants) | 98 | 100 | 96 | 86 | 98
  Arthralgia at Dose 1 | 20 | 15 | 9 | 9 | 18
  Fatigue at Dose 1: number analyzed (Participants) | 99 | 102 | 100 | 92 | 100
  Fatigue at Dose 1 | 56 | 61 | 55 | 46 | 50
  Nausea at Dose 1: number analyzed (Participants) | 97 | 101 | 97 | 85 | 99
  Nausea at Dose 1 | 16 | 23 | 14 | 13 | 14
  Headache at Dose 1: number analyzed (Participants) | 98 | 102 | 98 | 92 | 99
  Headache at Dose 1 | 40 | 46 | 38 | 36 | 36
  Myalgia at Dose 1: number analyzed (Participants) | 98 | 101 | 97 | 87 | 99
  Myalgia at Dose 1 | 34 | 29 | 27 | 21 | 28
  Fever at Dose 1: number analyzed (Participants) | 100 | 103 | 100 | 94 | 101
  Fever at Dose 1 | 6 | 5 | 5 | 1 | 3
  Arthralgia at Dose 2: number analyzed (Participants) | 98 | 103 | 98 | 92 | 0
  Arthralgia at Dose 2 | 22 | 19 | 12 | 17 |
  Fatigue at Dose 2: number analyzed (Participants) | 100 | 104 | 100 | 94 | 0
  Fatigue at Dose 2 | 58 | 61 | 62 | 56 |
  Nausea at Dose 2: number analyzed (Participants) | 98 | 102 | 98 | 93 | 0
  Nausea at Dose 2 | 16 | 13 | 15 | 17 |
  Headache at Dose 2: number analyzed (Participants) | 98 | 104 | 100 | 93 | 0
  Headache at Dose 2 | 52 | 36 | 37 | 39 |
  Myalgia at Dose 2: number analyzed (Participants) | 98 | 103 | 99 | 94 | 0
  Myalgia at Dose 2 | 41 | 38 | 35 | 38 |
  Fever at Dose 2: number analyzed (Participants) | 100 | 104 | 100 | 94 | 0
  Fever at Dose 2 | 6 | 3 | 3 | 1 |

13. Secondary Outcome: Number of Subjects With Unsolicited AEs
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e. lack of efficacy), abuse or misuse. An unsolicited AE is an AE that was not solicited using a Subject Diary and that was spontaneously communicated by a subjects/parent(s)/ Legally Acceptable Representative who has signed the informed consent or a solicited local or systemic adverse event that continues beyond the solicited period at day 7 after vaccination.
Time Frame: During the 30 days (including the day of vaccination) after each vaccination i.e after Dose 1 administered at Day 1 (for all groups) and after Dose 2 administered at Day 61 (for all groups except for MenACWY Group)
Population: Analysis was performed on unsolicited safety set that included all subjects who provided informed consent,underwent screening procedures,had a subject number assigned,received any study vaccination & was reported with any unsolicited AE data.No results for dose 2 category for subjects of MenACWY Group as they received only 1 dose at day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | MenABCWY Group | rMenBOMV+ACWY_S Group | rMenBOMV+ACWY_D Group | rMenBOMV Group | MenACWY Group
Number analyzed (Participants) | 100 | 104 | 100 | 94 | 102
Participants
  Any unsolicited AEs- Dose 1 | 16 | 19 | 16 | 16 | 15
  Any unsolicited AEs- Dose 2: number analyzed (Participants) | 100 | 104 | 100 | 94 | 0
  Any unsolicited AEs- Dose 2 | 11 | 14 | 13 | 10 |

14. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs), Medically Attended AEs (MAEs), AEs Leading to Withdrawal, and Adverse Events of Special Interest (AESIs)
Description: SAE is defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability or incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Medically attended AEs are defined as symptoms or illnesses requiring hospitalization, or emergency room visit, or visit to/by a health care provider. AESIs are predefined (serious or non-serious) adverse events of scientific and medical concern specific to the product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate, because such an event might warrant further investigation in order to characterize and understand it.
Time Frame: During the whole study period i.e from Day 1 to Day 91
Population: Analysis was performed on the unsolicited safety set that included all subjects who provided informed consent, underwent screening procedures, had a subject number assigned, received any study vaccination and was reported with any adverse event data.
Measure: Count of Participants; unit: Participants
Arm/Group | MenABCWY Group | rMenBOMV+ACWY_S Group | rMenBOMV+ACWY_D Group | rMenBOMV Group | MenACWY Group
Number analyzed (Participants) | 100 | 104 | 100 | 94 | 102
Participants
  SAE(s) | 0 | 2 | 1 | 2 | 0
  MAE(s) | 14 | 17 | 14 | 13 | 6
  AE(s) leading to withdrawal | 0 | 0 | 0 | 0 | 0
  AESI(s) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited Adverse Events were reported during the 7 days post-vaccination period and Unsolicited Adverse Events during the 30 Days post-vaccination period. Serious Adverse Events: were reported during the whole study period (from Day 1 up to Day 91).
Arm/Group | MenABCWY Group | rMenBOMV+ACWY_S Group | rMenBOMV+ACWY_D Group | rMenBOMV Group | MenACWY Group
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/104 | 0/100 | 0/94 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/100 | 2/104 | 1/100 | 2/94 | 0/102
Other Adverse Events (participants affected / at risk) | 94/100 | 103/104 | 98/100 | 94/94 | 80/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenABCWY Group (N=100) | rMenBOMV+ACWY_S Group (N=104) | rMenBOMV+ACWY_D Group (N=100) | rMenBOMV Group (N=94) | MenACWY Group (N=102)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenABCWY Group (N=100) | rMenBOMV+ACWY_S Group (N=104) | rMenBOMV+ACWY_D Group (N=100) | rMenBOMV Group (N=94) | MenACWY Group (N=102)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 3 (3) | 0 (0) | 3 (3) | 3 (3)
Viral infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 70 (114) | 74 (122) | 72 (117) | 63 (102) | 50 (50)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 24 (32) | 26 (36) | 26 (29) | 26 (30) | 14 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 (42) | 29 (34) | 18 (21) | 19 (26) | 18 (18)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericoronitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 50 (75) | 49 (67) | 45 (64) | 41 (59) | 28 (28)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Injection site pain (General disorders) | 94 (176) | 102 (197) | 97 (190) | 93 (175) | 53 (53)
Erythema (General disorders) | 50 (78) | 71 (108) | 57 (82) | 58 (81) | 28 (28)
Swelling (General disorders) | 51 (80) | 63 (98) | 46 (69) | 46 (65) | 23 (23)
Induration (General disorders) | 44 (65) | 54 (85) | 49 (72) | 38 (56) | 19 (19)
Pyrexia (General disorders) | 12 (13) | 7 (8) | 8 (8) | 2 (2) | 3 (3)
Injection site induration (General disorders) | 2 (2) | 5 (5) | 1 (1) | 4 (4) | 0 (0)
Injection site erythema (General disorders) | 2 (2) | 3 (3) | 4 (4) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 3 (4) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Vaccination site erythema (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Vaccination site swelling (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Vaccination site induration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site hypersensitivity (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site discolouration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 60 (92) | 57 (82) | 54 (75) | 52 (75) | 36 (36)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/07/NCT03587207/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT03587207/SAP_001.pdf